CLINICAL TRIAL: NCT02535923
Title: CBT-I for Psychosis: Guidelines, Preliminary Efficacy, and Functional Outcomes
Acronym: CBT-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Maryland Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D1836-W; 1IK2RX001836-01A1 (NIH)
Record Dates: First submitted 2015-08-26; First posted 2015-08-31 (Estimated); Results first posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Insomnia; Psychosis
Keywords: Schizophrenia and Disorders with Psychotic Feature; Mental Disorders; Insomnia Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Psychotic Disorders; Schizophrenia; Mental Disorders | interventions — Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Behavioral Therapy-Insomnia (Experimental): CBT-I addresses cognitive, arousal and behavioral factors related to sleep difficulties. Sessions combine assessment, conceptualization, psychoeducation, behavioral strategies and cognitive therapy, using a consistent structure including review of participants' sleep log and adherence to behavioral guidelines, modification of time in bed, cognitive therapy, and relaxation techniques. CBT-I also incorporates psychoeducation about biological and psychological elements that regulate sleep. Other strategies include stimulus control (i.e., getting out of bed when not sleepy) to extinguish the conditioned arousal common in insomnia, and relaxation techniques to reduce arousal associated with the bed, bedroom, or bedtime.
  Interventions: Behavioral: Cognitive Behavioral Therapy-Insomnia
- Health and Wellness (Active Comparator): Health and Wellness is a general self-management curriculum focused on providing education and support for managing physical and emotional well-being. Each session follows a basic structure including review of previous session material, new educational information and discussion on several topics over the course of single or multiple sessions. Each session will focus on the impact of the topic on overall health and wellness, identifying benefits and challenges to improving or maintaining health in that area, and strategies that clients may find helpful to address challenges in that area. Example topics include physical activity/exercise, nutrition/healthy eating, managing medications and side effects, and addictive behaviors (e.g., substance use, gambling, eating).
  Interventions: Behavioral: Health and Wellness

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy-Insomnia — CBT-I addresses cognitive, arousal and behavioral factors related to sleep difficulties. Sessions combine assessment, conceptualization, psychoeducation, behavioral strategies and cognitive therapy, using a consistent structure including review of participants' sleep log and adherence to behavioral guidelines, modification of time in bed, cognitive therapy, and relaxation techniques. CBT-I also incorporates psychoeducation about biological and psychological elements that regulate sleep. Other strategies include stimulus control (i.e., getting out of bed when not sleepy) to extinguish the conditioned arousal common in insomnia, and relaxation techniques to reduce arousal associated with the bed, bedroom, or bedtime.
  Arms: Cognitive Behavioral Therapy-Insomnia
Behavioral: Health and Wellness — Health and Wellness is a general self-management curriculum focused on providing education and support for managing physical and emotional well-being. Each session follows a basic structure including review of previous session material, new educational information and discussion on several topics over the course of single or multiple sessions. Each session will focus on the impact of the topic on overall health and wellness, identifying benefits and challenges to improving or maintaining health in that area, and strategies that clients may find helpful to address challenges in that area. Example topics include physical activity/exercise, nutrition/healthy eating, managing medications and side effects, and addictive behaviors (e.g., substance use, gambling, eating).
  Arms: Health and Wellness

SUMMARY:
The goal of this project is to develop guidelines for the clinical tailoring of Cognitive Behavioral Therapy for Insomnia (CBT-I) for Veterans with psychotic disorders and insomnia, and to test the acceptability, feasibility, and preliminary efficacy of CBT-I for improving sleep-related functional outcomes in this population.

DETAILED DESCRIPTION:
The goal of this project is to develop guidelines for the clinical tailoring of Cognitive Behavioral Therapy for Insomnia (CBT-I) for Veterans with psychotic disorders and insomnia, and to test the acceptability, feasibility, and preliminary efficacy of CBT-I for improving sleep-related functional outcomes in this population.

Specific Aim 1: Develop empirically-derived guidelines for the clinical tailoring of CBT-I materials and procedures for Veterans with psychotic disorders through an iterative process with input from Veteran clients, CBT-I experts and providers, as well as those with expertise in psychotic disorders.

Specific Aim 2: Establish the acceptability of CBT-I for Veterans with psychotic disorders and insomnia when delivered using guidelines developed in Specific Aim 1 in order to make further refinements to the guidelines in a preliminary trial with 6 Veterans with psychosis and insomnia.

Specific Aim 3: Conduct a randomized controlled trial (n=60) to test the feasibility and preliminary efficacy of CBT-I in producing positive changes at post-treatment and 3-month follow-up on the outcomes of insomnia symptoms, sleep quality, and functioning.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnostic and Statistical Manual of Disorders, 5th edition (DSM 5) diagnosis of schizophrenic disorders (295.0-295.9), affective psychoses (296.0-296.1, 296.4-296.8), or major depression with psychotic features (296.24, 296.34).
2. Self-reported symptoms of insomnia via an Insomnia Severity Index (ISI) score of 15 or greater.
3. Age between 18 and 80 as determined by medical record review.
4. Participation in outpatient mental health services at a designated study site.
5. Sufficient clinical stability to participate as deemed by a treatment provider.
6. Capacity to sign Informed Consent.

Exclusion Criteria:

1. Current problematic drug or alcohol use that impacts functioning and study engagement, as deemed by a treatment provider.
2. Currently in CBT-I treatment, determined by medical records.
3. Positive screen for sleep apnea via a portable sleep apnea screening device or a prior diagnosis of sleep apnea in medical records.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A. Klingaman, PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohrs S. Sleep disturbances in patients with schizophrenia : impact and effect of antipsychotics. CNS Drugs. 2008;22(11):939-62. doi: 10.2165/00023210-200822110-00004. PMID 18840034
- [Background] Bramoweth AD, Germain A. Deployment-related insomnia in military personnel and veterans. Curr Psychiatry Rep. 2013 Oct;15(10):401. doi: 10.1007/s11920-013-0401-4. PMID 24005883
- [Background] Klingaman EA, Palmer-Bacon J, Bennett ME, Rowland LM. Sleep Disorders Among People With Schizophrenia: Emerging Research. Curr Psychiatry Rep. 2015 Oct;17(10):79. doi: 10.1007/s11920-015-0616-7. PMID 26279058
- [Background] Buysse DJ. Insomnia. JAMA. 2013 Feb 20;309(7):706-16. doi: 10.1001/jama.2013.193. PMID 23423416
- [Background] Irwin MR, Cole JC, Nicassio PM. Comparative meta-analysis of behavioral interventions for insomnia and their efficacy in middle-aged adults and in older adults 55+ years of age. Health Psychol. 2006 Jan;25(1):3-14. doi: 10.1037/0278-6133.25.1.3. PMID 16448292
- [Background] Myers E, Startup H, Freeman D. Cognitive behavioural treatment of insomnia in individuals with persistent persecutory delusions: a pilot trial. J Behav Ther Exp Psychiatry. 2011 Sep;42(3):330-6. doi: 10.1016/j.jbtep.2011.02.004. Epub 2011 Mar 2. PMID 21367359
- [Background] Dopke CA, Lehner RK, Wells AM. Cognitive-behavioral group therapy for insomnia in individuals with serious mental illnesses: a preliminary evaluation. Psychiatr Rehabil J. 2004 Winter;27(3):235-42. doi: 10.2975/27.2004.235.242. PMID 14982330

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy-Insomnia | Health and Wellness
Started | 26 | 21
Completed Post Assessment | 22 (4 lost contact or refused) | 17 (4 lost contact or refused)
Completed Follow Up Assessment | 17 (5 lost contact or refused) | 13 (4 lost contact or refused)
Completed | 17 | 13
Not Completed | 9 | 8
Not completed — Lost to Follow-up | 5 | 5
Not completed — Withdrawal by Subject | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Therapy-Insomnia | Health and Wellness | Total
Number analyzed (Participants) | 26 | 21 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (10.6) | 50.4 (12.6) | 51.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 19 | 17 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 11 | 19
  White | 15 | 6 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7
Insomnia Severity Index [Mean (Standard Deviation); unit: units on a scale] — Scale ranges from 0-28, with higher scores indicating more severe insomnia.
  units on a scale | 18.7 (5.1) | 18.1 (5.6) | 18.5 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity Index (ISI)
Description: ISI score; scored on a scale of 0 to 28, with higher scores indicating worse insomnia severity.
Time Frame: Participants will be assessed following completion of the study intervention, an expected average of 10 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy-Insomnia | Health and Wellness
Number analyzed (Participants) | 22 | 17
units on a scale | 11.6 (7.5) | 15.2 (4.5)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy-Insomnia vs Health and Wellness; Test type: Superiority; p = .04, Mixed Models Analysis
Statistical Analysis 2: Comparison: Cognitive Behavioral Therapy-Insomnia vs Health and Wellness; Test type: Superiority; p = .83, Mixed Models Analysis

2. Secondary Outcome: Insomnia Severity Index (ISI)
Description: ISI score; scored on a scale of 0 to 28, with higher scores indicating worse insomnia severity.
Time Frame: Participants will be assessed a second time following completion of the study intervention, an expected average of 22 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy-Insomnia | Health and Wellness
Number analyzed (Participants) | 17 | 13
units on a scale | 12.4 (7.4) | 13.0 (6.0)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy-Insomnia vs Health and Wellness; Test type: Superiority; p = .83, Mixed Models Analysis

3. Secondary Outcome: Veterans RAND 36-Item Health Survey Mental Component Score
Description: Veterans RAND 36-Item Health Survey score Mental Component Score; Possible scores range from 0 to 100, with higher scores indicating greater mental quality of life.
Time Frame: Participants will be assessed following completion of the study intervention, an expected average of 10 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy-Insomnia | Health and Wellness
Number analyzed (Participants) | 22 | 17
units on a scale | 40.0 (13.8) | 45.5 (10.8)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy-Insomnia vs Health and Wellness; Test type: Superiority; p = .003, Mixed Models Analysis

4. Secondary Outcome: Veterans RAND 36-Item Health Survey Mental Component Score
Description: Veterans RAND 36-Item Health Survey Mental Component Score; Possible scores range from 0 to 100, with higher scores indicating greater mental health quality of life.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy-Insomnia | Health and Wellness
Number analyzed (Participants) | 17 | 13
units on a scale | 48.4 (12.2) | 47.8 (12.6)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy-Insomnia vs Health and Wellness; Test type: Superiority; p = .16, Mixed Models Analysis

5. Secondary Outcome: World Health Organization Disability Assessment Schedule (WHO-DAS), Participation in Society Subscale
Description: WHO-DAS score; scores range from 0 to 100 where 100 is full disability.
Time Frame: Participants will be assessed following completion of the study intervention, an expected average of 10 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy-Insomnia | Health and Wellness
Number analyzed (Participants) | 22 | 17
units on a scale | 39.9 (22.3) | 34.1 (25.8)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy-Insomnia vs Health and Wellness; Test type: Superiority; p = .82, Mixed Models Analysis

6. Secondary Outcome: World Health Organization Disability Assessment Schedule (WHO-DAS), Participation in Society Subscale
Description: WHO-DAS score; scores range from 0 to 100 where 100 is full disability.
Time Frame: Participants will be assessed a second time following completion of study intervention, an estimated average of 22 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy-Insomnia | Health and Wellness
Number analyzed (Participants) | 17 | 13
units on a scale | 42.9 (22.7) | 29.6 (15.6)

ADVERSE EVENTS:
Time Frame: From baseline to an average of 22 weeks per participant.
Arm/Group | Cognitive Behavioral Therapy-Insomnia | Health and Wellness
All-Cause Mortality (participants affected / at risk) | 2/26 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/21
Other Adverse Events (participants affected / at risk) | 1/26 | 0/21
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Behavioral Therapy-Insomnia (N=26) | Health and Wellness (N=21)
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — A participant wore a watch device according to the protocol and experienced skin irritation where the device was worn.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/23/NCT02535923/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-27): https://cdn.clinicaltrials.gov/large-docs/23/NCT02535923/ICF_001.pdf